CLINICAL TRIAL: NCT06235307
Title: Effects of Motivational Interviewing on Compliance With Physical Activity Practice in Patients With Chronic Disease in the City of Amiens
Brief Title: Motivational Interviewing and Practice of Physical Activity in Patients With ALD
Acronym: MOTIVAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2023_843_0092
Record Dates: First submitted 2024-01-09; First posted 2024-01-31 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Motivational Interviewing; Chronic Disease
Keywords: motivational interviewing; physical activity practice; Chronic Disease; IPAQ score; SF12 score
MeSH Terms: conditions — Chronic Disease | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- motivational interviewing (Experimental)
  Interventions: Other: motivational interviewing
- Control (Active Comparator)
  Interventions: Other: motivational interviewing

INTERVENTIONS:
Other: motivational interviewing — Upon entry into the program, all patients will be seen for an assessment of their physical condition at the premises of Amiens Métropole by a teacher in adapted physical activity (APA) in order to be assessed and directed to a club or a approved associations. The EM group will also benefit from a motivational interview at 0 and 3 months by a doctor trained in the technique. The entire cohort will complete the SF12 (perception of quality of life) and IPAQ (current level of physical activity) questionnaires at 0 and 6 months during the usual appointments with the APA teacher.

SUMMARY:
Since 2017, ALD patients can be prescribed Adapted Physical Activity (APA) on prescription. However, this possibility of prescription remains relatively unknown and little used by doctors, while the benefits of APA in particular in chronic diseases are well established and 30% of adults in France do not reach the recommendations of WHO on physical activity. These obstacles to prescription are well known thanks to studies on the subject (lack of information on Sport-Health networks, lack of training in APA prescription, poor financial support, lack of support for deliver to patients).

To overcome this lack of implementation, the city of Amiens, via the Office des Sports d'Amiens Métropole (OSAM), has implemented since September 2022 tools to help prescribe APA: blocks pre- filled certificates of absence of contraindication and prescription of adapted physical activity.

In other areas of health, such as breastfeeding, performing motivational interviewing has improved patient compliance. Patients with chronical disease consult a doctor from the Amiens metropolitan area recruited beforehand who informs them of the existence of the physical activity promotion program of Amiens Métropole. After obtaining their consent and establishing a certificate of no contraindication, the patients will be randomized by a random draw into two groups: motivational interviewing (ME) and control group (GT). Upon entry into the program, all patients will be seen for an assessment of their physical condition at the premises of Amiens Métropole by a teacher in adapted physical activity (APA) in order to be assessed and directed to a club or a approved associations. The EM group will also benefit from a motivational interview at 0 and 3 months by a doctor trained in the technique. The entire cohort will complete the SF12 (perception of quality of life) and IPAQ (current level of physical activity) questionnaires at 0 and 6 months during the usual appointments with the APA teacher.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic disease (ALD)
* aged 18 and over, autonomous in their ability to move
* living in the metropolis of Amiens

Exclusion Criteria:

* contraindication to the practice of physical activity;
* patient under guardianship, curators,
* safeguard of justice ;
* patient deprived of liberty ;
* pregnant woman ;
* patient who not benefiting from a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
change from baseline of the IPAQ score | 3 months
  IPAQ is the International Physical Activity Questionnaire Measurement of the evolution of the IPAQ score of patients according to participation in motivational interviewing

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire d'Amiens, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No